CLINICAL TRIAL: NCT05329883
Title: Multicentric Study on Infections of the Urinary Tract After Stent Removal (MINUS-trial).
Acronym: MINUS
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Collaborators: AZ Sint-Lucas Gent (Other); Universitaire Ziekenhuizen KU Leuven (Other); General Hospital Groeninge (Other); University of British Columbia (Other); Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Other Study IDs: BC-10846
Record Dates: First submitted 2022-03-25; First posted 2022-04-15 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Urinary Tract Infections; Stent Related Infection
Keywords: Urinary Tract Infection; Ureteral stent removal; Double-J stent; Ureterorenoscopy; Percutaneous Nephrolithotomy; Endourology
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Weeks
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: Double-J stent removal — Outpatient ureteral stent removal without antibiotic prophylaxis

SUMMARY:
The MINUS-trial is a multicentric prospective observational study in which consecutive patients, 18 years of age and older who receive a ureteral stent during any endoscopic procedure will be approached to participate. Their stent will be removed in outpatient office or by string extraction at home with or without antibiotic prophylaxis (depending on the standard of care of the participating center). A urine sample will be taken before stent removal and patients will be asked to complete a questionnaire to assess symptoms of urinary tract infection (UTI) after stent removal. If the patient experiences symptoms of UTI (urgency, frequency, dysuria or haematuria) that exceed the usually experienced post-cystoscopy symptoms, they have to provide a urine sample.

The purpose of this study is to provide multi-institutional, multinational, observational data on the incidence of UTI after stent removal with or without antibiotic prophylaxis in the outpatient setting in patients with a sterile urine culture prior to the intervention of stent placement and no demonstrated infection during the stent has been in situ.

The primary outcome is the presence of a febrile or non-febrile urinary tract infection after stent removal.

Secondary objectives are to identify risk factors for post-stent removal UTI and identify differences in UTI incidence between cystoscopic stent removal in the outpatient setting versus string-removal by the patient in the home environment.

DETAILED DESCRIPTION:
Given the high morbidity, cost and loss of quality of life of stent related infections, there is a need for practical strategies for decreasing stent associated UTI's and sepsis. One of these strategies may be to provide targeted antibiotic prophylaxis. On the other hand, the widespread growing bacterial resistance due to the overuse of antibiotics is of growing concern.

To date, no clear guidelines regarding antibiotic prophylaxis prior to ureteral stent removal are available. The European Association of Urology (EAU) does not recommend antibiotic prophylaxis before cystoscopy, but there is no specific recommendation regarding stent removal. This is mainly due to the lack of good and robust data.

The MINUS-trial is a multicentric prospective observational study with the aim of providing multi-institutional, multinational, observational data on the incidence of UTI after stent removal with or without antibiotic prophylaxis in the outpatient setting in patients with a sterile urine culture prior to the intervention of stent placement and no demonstrated infection during the stent has been in situ.

The primary outcome is the presence of a febrile or non-febrile urinary tract infection after stent removal.

Secondary objectives are to identify risk factors for post-stent removal UTI and identify differences in UTI incidence between cystoscopic stent removal in the outpatient setting versus string-removal by the patient in the home environment.

All consecutive patients, 18 years of age and older who receive a ureteral stent during any endoscopic procedure will be approached to participate. Their stent will be removed in outpatient office or by string extraction at home with or without antibiotic prophylaxis (depending on the standard of care of the participating center). A urine sample will be taken before stent removal and patients will be asked to complete a questionnaire to assess symptoms of urinary tract infection (UTI) after stent removal. If the patient experiences symptoms of UTI (urgency, frequency, dysuria or haematuria) that exceed the usually experienced post-cystoscopy symptoms, they have to provide a urine sample.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 years or above
* Stent placed during endoscopic procedure
* A negative urine culture (UC) pre-operatively with a single dose of antibiotic prophylaxis peri-operatively
* Stent removal is planned in outpatient setting of by the patient by using a string.
* Able and willing to provide consent

Exclusion Criteria:

* Permanent indwelling catheter (transurethral catheter, suprapubic catheter, nephrostomy tubes)
* Pregnant patients
* Patient performing clean intermittent (self-)catheterization
* Recent history (<3 months) of demonstrated UTI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients, 18 years of age and older who receive a ureteral stent during any endoscopic procedure will be approached to participate in the study
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-11-25 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
number of participants demonstrating a post-stent removal urinary tract infection | 30 days after removal
  For this outcome measure, a urinary tract infection is defined as a urine sample demonstrating an identified uropathogen with at least 10.000 colony forming units in a patient demonstrating symptoms of a urinary tract infection after removal of a ureteral stent. Asymptomatic bacteriuria will not be considered a positive outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Ghent, Ghent, Eastern-Flanders, Belgium

IPD SHARING:
Plan to Share IPD: No